CLINICAL TRIAL: NCT04412239
Title: To Assess the Efficiency and Satisfaction of Pharmacist Giving Patient-centred Advice on Telephone Consultation in TB Patients: Experience of the COVID-19 Pandemic
Acronym: Coronavirus19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xi'an Jiaotong University (Other)
Collaborators: Pakistan Institute of Medical Sciences (Other Government); District Headquarter Hospital Bannu Pakistan (Unknown)
Responsible Party: Principal Investigator, Farman Ullah Khan, Department of Pharmacy Administration and Clinical Pharmacy School of Pharmacy, Health Science Centre Xi'an Jiao tong University., Xi'an Jiaotong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NO, F6-2017/NTP-ADMIN
Record Dates: First submitted 2020-05-30; First posted 2020-06-02 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: TB - Tuberculosis; Patient Satisfaction
MeSH Terms: conditions — Latent Tuberculosis; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telephone Consultation in TB Patients (Experimental): The COVID-19 pandemic might be an opportunity to review and refine our practices in TB care. For the follow-up of selected patients, telephone consultations may be efficient and cost-effective.
  Interventions: Behavioral: Patient-centred advice on Telephone Consultation in TB Patients:

INTERVENTIONS:
Behavioral: Patient-centred advice on Telephone Consultation in TB Patients: — The primary aim was to assess the efficiency and the satisfaction of the telephone consultation. The COVID-19 pandemic might be an opportunity to review and refine our practices in TB care. For the follow-up of selected patients, telephone consultations may be efficient and cost effective.

SUMMARY:
The COVID-19 pandemic might be an opportunity to review and refine our practices in anti TB treatment. For the follow-up of selected patients, telephone consultations may be efficient and cost-effective. The aim of the study is to assess the efficiency and the satisfaction with telephone consultation for the pharmacist and the TB patient. The study was conducted in tertiary care hospital TB control centres patients.

DETAILED DESCRIPTION:
Tuberculosis (TB) is the world's biggest killer among infectious diseases, claiming more than 4000 lives each day. The unprecedented coronavirus pandemic seriously impacts people with pre-existing health conditions. People who have TB are usually more vulnerable to other infections, including the novel coronavirus, due to pre-existing lung damage. They are at a higher risk of developing complications from COVID-19. Certain populations are at greater risk of TB, because of where they live, where they work or because of other socio-economic factors which result in them experiencing barriers to accessing health services.

ELIGIBILITY:
Inclusion Criteria:

New, smear-positive drug-susceptible TB who have been on treatment for less than two weeks Access to a mobile phone (self-reported)

Exclusion Criteria:

Patients who do not have regular access to a mobile phone Patients who have previously received TB treatment Patients who have another member in their household who is already a part of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-12-20 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Efficiency of the telephone consultation, | 2 Months
  To improve patient centered care/patient prescription refill
Patient satisfaction | 2 Month
  Patient satisfaction Patient satisfaction resulting from pharmacist-led pharmaceutical care will be assessed Patient satisfaction feedback (PSF)

SECONDARY OUTCOMES:
Adherence Rate | 2 Months

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Dhq Bannu Kpk, Bannu, KPK
  - District Bannu TB Control Center, Bannu, KPK